CLINICAL TRIAL: NCT02020057
Title: Comparison of Highly Cross-Linked and Conventional Polyethylene in Posterior Cruciate-Substituting Total Knee Arthroplasty in the Same Patients
Brief Title: Comparison of Highly Cross-Linked and Conventional Polyethylene in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSXL; 2006-32 (Other: Institutional Review Board, Dongdaemun Hospital)
Record Dates: First submitted 2013-12-13; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): knee receiving Total knee arthroplasty with conventional polyethylene inserts
  Interventions: Procedure: Total knee arthroplasty
- Prolong (Experimental): knee receiving total knee arthroplasty with highly cross linked polyethylene insert
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty with standard incision and approach, and cement fixation. Zimmer Nexgen posterior stabilized total knee implants are used.

SUMMARY:
To our knowledge, there has been no information on in vivo clinical results of posterior cruciate-substituting arthroplasties using highly cross-linked polyethylene. We evaluated whether the clinical and radiographic results, incidence of post fracture of the tibial polyethylene insert, failure of the locking mechanism of the tibial polyethylene insert, and the incidence of osteolysis would be similar between posterior cruciate-substituting total knee prostheses using conventional and highly cross-linked polyethylene.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis that was severe enough to warrant total knee arthroplasty after an adequate trial of nonoperative therapy, and the need for bilateral total knee arthroplasties

Exclusion Criteria:

* inflammatory arthritis
* osteoarthritis of the hip causing pain or restricted mobility
* a foot or ankle disorder which limited walking
* dementia or a neurological disorder including a past history of stroke which affected mobility

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-02; Primary Completion 2010-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
knee society knee score | 3 months, 1 year, and yearly thereafter the operation, until 15 years after the operation
  clinical evaluation of knee function by knee score. This knee score will be compared, between preoperative and the latest score, and between the latest scores of study and control group.

SECONDARY OUTCOMES:
range of motion | preoperative, 3 months, 1 year, and yearly thereafter the operation until 15 years
  this value will be compared between preoperative and the latest value, and between the latest value of study and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, M.D., Study Director — Ewha Womans University Mokdong Hospital